CLINICAL TRIAL: NCT02128035
Title: Radiation Protection With a Pelvic Lead Shield and a Radiation Protection Cap for Operators Performing Coronary Angiography or Intervention, a Randomized Controlled Trial
Brief Title: RADIATION PROTECTion With a Pelvic Lead Shield and a Radiation Protection Cap for Operators Performing Coronary Angiography or Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sanjit S. Jolly (Other)
Collaborators: McMaster University (Other); Population Health Research Institute (Other)
Responsible Party: Sponsor-Investigator, Dr. Sanjit S. Jolly, Interventional Cardiologist, Associate Professor, Population Health Research Institute
Organization: Population Health Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RADIATION PROTECT; Project Number 12-520 (Other: Hamilton Health Sciences Research Ethics Board)
Record Dates: First submitted 2012-12-20; First posted 2014-05-01 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Acute Coronary Syndromes
Keywords: radiation protection; interventional cardiologist; percutaneous coronary intervention (PCI); angiography; lead shield
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Without Lead Shield (No Intervention): All routine measures to reduce radiation exposure (including lead aprons, lead collar, lead lenses, movable ceiling suspended lead shield with a long lead skirt attached to its lower margin) will be used as done routinely and will be left to the operators' discretion.
  The LEAD SHIELD will not be used in this group.
  Interventional cardiologists who will perform the procedure will wear a radiation protection cap in all procedures.
- With Lead Shield (Experimental): All routine measures to reduce radiation exposure (including lead aprons, lead collar, lead lenses, movable ceiling suspended lead shield with a long lead skirt attached to its lower margin) will be used as done routinely and will be left to the operators' discretion.
  In this group, a LEAD SHIELD will be used. The Pelvic lead shield will be draped on patient from umbilicus to knees.
  Interventional cardiologists who will perform the procedure will wear a radiation protection cap in all procedures.
  Interventions: Procedure: With Lead Shield

INTERVENTIONS:
Procedure: With Lead Shield — A pelvic lead shield will be draped on patient from umbilicus to knees.
  Interventional cardiologists who will perform the procedure will wear a radiation protection cap in all procedures.
  Arms: With Lead Shield

SUMMARY:
RADIATION PROTECT is a randomized, controlled trial of patients undergoing coronary angiography or PCI with or without a pelvic lead shield. Interventional cardiologists who will perform the procedure will wear a radiation protection cap in all procedures.

It is hypothesized that routine use of the pelvic lead shield and radiation protection cap during these procedures will reduce the amount of radiation in which the interventional cardiologists get exposed.

DETAILED DESCRIPTION:
Patients referred for coronary angiography or PCI will be randomized to undergo their procedure with or without the pelvic lead shield and the operator will wear a radiation protection cap.

Clinical efficacy will be assessed based on the total radiation dose that the interventional cardiologist got exposed to as well as a secondary outcome measuring the total radiation exposure dose per minute.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for coronary angiography or Percutaneous Coronary Intervention (PCI)

Exclusion Criteria:

* Age ≤ 18 years
* Previous inclusion in RADIATION PROTECT trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Total Radiation Dose | Duration of Procedure (an expected average of 30 minutes)
  1. The total radiation dose that the interventional cardiologist got exposed to as read by dosimeters (µSv) at left breast.
  2. The difference between both groups in radiation dose that the interventional cardiologist got exposed to divided by Air Kerma (µSv/mGy).
  3. For the radiation protection cap, the primary outcome is the difference between total radiation dose as measured by two dosimeters (µSv) at left temporal region of the head of the interventional cardiologist (one on the outside of the radiation protection cap and the other one on the inside of the cap).

SECONDARY OUTCOMES:
Radiation Exposure Dose per minute | Duration of Procedure (an expected average of 30 minutes)
  The difference between both groups in radiation exposure dose per minute (µSv /min) at left breast and left temporal region.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjit S Jolly, MD, Principal Investigator — Hamilton Health Sciences, McMaster University; Ashraf Al Azzoni, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Alazzoni A, Gordon CL, Syed J, Natarajan MK, Rokoss M, Schwalm JD, Mehta SR, Sheth T, Valettas N, Velianou J, Pandie S, Al Khdair D, Tsang M, Meeks B, Colbran K, Waller E, Fu Lee S, Marsden T, Jolly SS. Randomized Controlled Trial of Radiation Protection With a Patient Lead Shield and a Novel, Nonlead Surgical Cap for Operators Performing Coronary Angiography or Intervention. Circ Cardiovasc Interv. 2015 Aug;8(8):e002384. doi: 10.1161/CIRCINTERVENTIONS.115.002384. PMID 26253734